CLINICAL TRIAL: NCT01999738
Title: A Phase I A/B Study of the Folic Acid-Tubulysin Conjugate EC1456 In Patients With Advanced Solid Tumors
Brief Title: Folic Acid-Tubulysin Conjugate EC1456 In Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC1456-01
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Solid Tumors; Non Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A - MTD (Treatment 1) (Experimental): Treatment 1 is BIW on Days 1, 4, 8, and 11 of a 3-week schedule (BIW).
  Intervention: EC1456 and EC20
  Interventions: Drug: EC1456 and EC20
- Part A - MTD (Treatment 2) (Experimental): Treatment 2 is EC1456 QW on Days 1 and 8 of a 3-week schedule (QW).
  Intervention: EC1456 and EC20
  Interventions: Drug: EC1456 and EC20
- Part A - MTD (Treatment 3) (Experimental): Treatment 3 is EC1456 QW on Days 1, 8, and 15 of a 3-week schedule (CWD).
  Intervention: EC1456 and EC20
  Interventions: Drug: EC1456 and EC20
- Part A - MTD (Treatment 4) (Experimental): Treatment 4 is EC1456 QIW on Days 1, 2, 3, 4, 8, 9, 10, and 11 of a 3-week schedule (QIW).
  Intervention: EC1456 and EC20
  Interventions: Drug: EC1456 and EC20
- Part B - Efficacy (Treatment 5) (Experimental): Treatment 5 is EC1456 BIW. Once a dose is determined in Part A, Part B will begin with 3-6 subjects who will receive consecutive day dosing on Days 1, 2, 8, and 9 of a 3-week schedule. If this is not tolerated, the BIW cohort will continue with dosing on Days 1, 4, 8, and 11 of a 3-week schedule.
  Intervention: EC1456 and EC20
  Interventions: Drug: EC1456 and EC20
- Part B - Efficacy (Treatment 6) (Experimental): Treatment 6 is EC1456 QW on Days 1 and 8 of a 3-week schedule or CWD on Days 1, 8 and 15 of a 3-week schedule.
  Intervention: EC1456 and EC20
  Interventions: Drug: EC1456 and EC20
- Part B - Efficacy (Treatment 7) (Experimental): Treatment 7 is EC1456 QIW on Days 1, 2, 3, 4, 8, 9, 10, and 11 of a 3-week schedule for at least two cycles. If the patient is eligible to continue treatment (based upon treatment response and tolerability), he/she may opt to continue on the QIW schedule or change to the Treatment 6 regimen schedule (once its MTD and schedule have been determined).
  Intervention: EC1456 and EC20
  Interventions: Drug: EC1456 and EC20

INTERVENTIONS:
Drug: EC1456 and EC20 — EC1456 is small molecule drug conjugate of folic acid and tubulysin B hydrazide (TubBH) that specifically binds to the membrane-bound FR and gains entry into the cell via endocytosis.
  EC20 is Etarfolatide, a conjugate of folic acid and a tripeptide moiety that can efficiently chelate the radioisotope 99mTechnetium (99mTc). When etarfolatide is labeled with 99mTc, the product (99mTc-etarfolatide) is able to quantify FR expressing tissues with SPECT imaging.
  Other Names: Folic acid and tubulysin B hydrazide and etarfolatide

SUMMARY:
Phase 1A/B, multicenter, open-label, non-randomized, dose-escalation oncology study to evaluate the administration of EC1456 in advanced solid tumors. In part A, EC1456 will be dose escalated on 4 concurrently enrolling schedules. FR-positive expression on a 99mTc-etarfolatide scan is not required for inclusion in Part A.

Part B of the study will confirm the maximum tolerated dose (MTD) and the recommended Phase 2 (RP2) dose of EC1456, and evaluate the efficacy of EC1456 in NSCLC all subtype patient populations with FR-positive cancer in up to three schedules (i.e., twice weekly, once weekly, and four times weekly). FR-positive expression on a 99mTc-etarfolatide scan is required for inclusion in Part B.

Minimum length of patient participation is anticipated to be 10 weeks (two 3-week cycles followed by a 30 day follow-up period).

DETAILED DESCRIPTION:
In part A, EC1456 will be dose escalated on 4 concurrently enrolling schedules.

Treatment 1 is EC1456 BIW on Days 1, 4, 8, and 11 of a 3-week schedule (BIW); Treatment 2 is EC1456 QW on Days 1 and 8 of a 3-week schedule (QW); Treatment 3 is EC1456 QW on Days 1, 8, and 15 of a 3-week schedule (CWD) and Treatment 4 is EC1456 QIW on Days 1, 2, 3, 4, 8, 9, 10, and 11 of a 3-week schedule (QIW).

In part B, EC1456 will be dosed on 3 concurrently enrolling schedules:

Treatment 5 is EC1456 BIW. Once a dose is determined in Part A, Part B will begin with 3-6 subjects who will receive consecutive day dosing on Days 1, 2, 8, and 9 of a 3-week schedule. If this is not tolerated, the BIW cohort will continue with dosing on Days 1, 4, 8, and 11 of a 3-week schedule; Treatment 6 is EC1456 QW on Days 1 and 8 of a 3-week schedule or CWD on Days 1, 8 and 15 of a 3-week schedule; Treatment 7 is EC1456 QIW on Days 1, 2, 3, 4, 8, 9, 10, and 11 of a 3-week schedule for at least two cycles. If the patient is eligible to continue treatment (based upon treatment response and tolerability), he/she may opt to continue on the QIW schedule or change to the Treatment 6 regimen schedule (once its MTD and schedule have been determined).

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in Part A must receive the 99mTc- etarfolatide scan but they do not need to have FR-positive target lesions.

Parts A and B:

To qualify for enrollment, the following criteria must be met:

1. Patient must have the ability to understand and sign an approved informed consent form (ICF).
2. Patient must be ≥ 18 years of age.
3. Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Patient must have a life expectancy of > 3 months.
5. Patient must have at least one measurable lesion per RECIST v1.1 Criteria as assessed on baseline radiologic evaluation obtained no more than 28 days prior to beginning study therapy.
6. Patients with central nervous system (CNS) metastases that are symptomatic must have received therapy (e.g., surgery, XRT, gamma knife, etc.) and be neurologically stable and off of steroids. The patient should be off steroids at least 14 days before registration. Patients with asymptomatic CNS metastatic disease without associated edema, shift, and a requirement for steroids or anti-seizure medications may be eligible after discussion with the sponsor medical monitor.
7. Patients must have formalin fixed tissue (biopsy or FNA) available.
8. Patient must have recovered (to baseline/stabilization) from prior chemo or radio therapy and associated acute toxicities must have resolved to a NCI CTCAE V4 Grade 1 or less, with the exception of alopecia.
9. Patients treated with prior radiation therapy may be eligible if:

   1. Radiotherapy was completed at least 2 weeks before first dose of EC1456 and
   2. Patient has recovered from acute radiation toxicity.
10. Patients must have adequate organ function:

    1. Bone marrow reserve: Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; Platelets ≥ 100 x 109/L; Hemoglobin ≥ 9 g/dL.
    2. Cardiac:

    i. QTcFridericia (QTcF) < 450 msec on at least 2 of 3 screening ECG's. On site determination of QTcF may be used for screening purposes.

    ii. Left ventricular ejection fraction (LVEF) equal to or greater than the institutional lower limit of normal. LVEF must be evaluated within 28 days prior to C1D1.

    iii. Cardiac Troponin I or T within normal limit. (whichever troponin is done for screening will need to be done throughout the rest of the study).

    c. Hepatic: Total bilirubin ≤ 1.5 x the upper limit of normal (ULN); Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 3.0 x ULN OR ≤ 5.0 x ULN for patients with liver metastases.

    d. Renal: Serum creatinine ≤ 1.5 x ULN or for patients with serum creatinine > 1.5 ULN, creatinine clearance ≥ 50 mL/min.

    Patients of childbearing potential:
11. All women of childbearing potential MUST have a negative urine or serum pregnancy test within 1 week prior to the 99mTc-etarfolatide imaging procedure and within 1 week prior to treatment with EC1456.
12. Women of child bearing potential must practice an effective method of birth control (i.e., oral, transdermal or injectable contraceptives, intrauterine device [IUD], or double-barrier contraception, such as diaphragm and spermicidal jelly) for the duration of their participation in the trial through 90 days following the last dose of EC1456.
13. Male patients who are sexually active must practice an effective method of birth control (e.g., condom and spermicidal jelly) for the duration of their participation in the trial through 90 days following the last dose of EC1456.

    Patient and Disease Specific Inclusion Criteria: Part A

    EC1456 dose escalation cohorts (Treatments 1, 2, 3, and 4):
14. Patients must have pathologically confirmed metastatic or locally advanced solid cancer (preferably TNBC, NSCLC, ovarian, or endometrial cancers due to frequent high FR expression in these cancers) that has failed to respond to standard therapy, is not amenable to standard therapy, or for which standard therapy does not exist.
15. TNBC and ovarian patients must agree to submit results of BRCA 1/2 status (i.e., deleterious mutation present, mutation of unknown significance, no mutation detected) if known. BRCA testing is not required for study inclusion.
16. Patients must have received ≤ 4 prior lines of systemic anti-cancer therapy (including but not limited to cytotoxic agents, targeted inhibitors, and monoclonal antibodies). Hormonal therapies are not included toward this criterion.
17. Patients must undergo a 99mTc-etarfolatide SPECT imaging procedure in compliance with the Investigator's Imaging Operations Manual (IIOM). FR expression on 99mTc -etarfolatide SPECT is not required for inclusion in Treatments 1, 2, 3, and 4.

    (Patients who underwent a 99mTc-etarfolatide SPECT/CT imaging procedure as a subject on Endocyte study EC20.12 will not be required to have a repeat scan for participation in study EC1456-01 if the scan was obtained within 4 weeks of cycle 1 day 1 of EC1456 administration and has been deemed acceptable by Endocyte Imaging.)

    Part B Only:

    Patient and Disease Specific Inclusion Criteria: Part B

    Patients with FR-positive NSCLC (all subtypes): (Treatments 5, 6, and 7)
18. Patients with NSCLC (all subtypes) must have received one prior platinum based therapy for advanced or metastatic disease. No additional cytotoxic therapy for advanced or metastatic disease is allowed. Any number of prior targeted therapies (e.g., inhibitors of ALK, EGFR, and PD-1 or PD-L1) are allowed. Patients with known relevant genomic tumor aberrations (i.e., EGFR, ALK, ROS-1, etc) must have received and progressed on approved therapy for these aberrations. This information must be documented prior to study entry.
19. Patients must undergo a 99mTc-etarfolatide SPECT imaging procedure in compliance with the Investigator's Imaging Operations Manual (IIOM) and be FR-positive.

Exclusion Criteria:

Parts A and B:

The presence of any of the following will exclude patients from the study:

1. Systemic anti-cancer treatment, except hormonal treatment, within 28 days prior to EC1456 administration unless there are no remaining or ongoing uncontrolled toxicities. Please contact the medical monitor to discuss requests for less than 28 day washout period.
2. Known hypersensitivity to the components of the study therapy or its analogs.
3. Carcinomatous meningitis and/or symptomatic central nervous system (CNS) metastases.
4. Malignancies that are expected to alter life expectancy or may interfere with disease assessment. Patients with adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, or low-grade (Gleason score ≤ 6) localized prostate cancer, ductal carcinoma in situ (DCIS), and patients with prior history of malignancy who have been disease free for more than 3 years are eligible.
5. Serious cardiac illness or medical conditions such as unstable angina, pulmonary embolism, or uncontrolled hypertension.
6. Patients considered at risk for life-threatening QTc prolongation (i.e., personal or family history of Long QT syndrome, presence of implantable pacemaker or implantable cardioverter defibrillator, etc.).
7. Use of the following medications within 6 months prior to EC1456 administration: amiodarone, disopyramide, dofetilide, dronedarone, flecanamide, ibutilide, quinidine, or sotalol.
8. Need for concurrent anti-folate therapy such as methotrexate for rheumatoid arthritis.
9. Other concurrent chemotherapy, immunotherapy, radiotherapy, or investigational therapy.
10. Pregnant or lactating women.
11. Active uncontrolled infections.
12. Known active Hepatitis B or C infection.
13. Unable or unwilling to have a pretreatment scan performed with 99mTc-etarfolatide for any reason (such as claustrophobia, an inability to lie supine on an imaging table because of pain or cardiopulmonary disease, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2) - Part A | 18-24 months
  Part A - To dose escalate EC1456 dose until maximum tolerated dose (MTD) and recommended Phase 2 (RP2) dose for multiple schedules is reached.
  -All patients who receive at least one dose of EC1456 will be evaluated for safety. All AEs and SAEs will be graded as per CTCAE V4.0. For each dose level, summaries of dose adjustments, adverse event rates, laboratory changes, cumulative toxicity, and dose limiting toxicity (DLT) will be analyzed. Summaries of CTCAE grades will be analyzed at each dose level and each cycle.
Efficacy Analysis - Part B | 18-24 months
  Part B - Response to study therapy will be calculated per RECIST v1.1 criteria for all patients treated with at least one dose of EC1456

CONTACTS AND LOCATIONS:
Overall Officials: Alison Armour, MD, Study Director — Endocyte
Locations (16):
- United States (16):
  - Mayo Clinic, Phoenix, Arizona
  - Honor Health, Scottsdale, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope, Duarte, California
  - Northwestern University Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - IU Health Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Horizon BioAdvance, Lafayette, Indiana
  - University of Maryland-Greenebaum Cancer Center, Baltimore, Maryland
  - Henry Ford Hospital - Josephine Ford Cancer Center, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - University Hospitals Case Medical Center - Seidman Cancer Center, Cleveland, Ohio
  - Westchase Clinical Associates, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Vermont Cancer Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No